CLINICAL TRIAL: NCT02096497
Title: In Vivo Analysis of the Vascular Pattern of the Superficial Temporal Artery Based on Digital Subtraction Angiography
Brief Title: Analysis of the Vascular Pattern of the Superficial Temporal Artery
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: BGU-001
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Arteria Temporalis Superficialis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (11):
- Vascular pattern 1
- Vascular pattern 2
- Vascular pattern 3
- Vascular pattern 4
- Vascular pattern 5
- Vascular pattern 6
- Vascular pattern 7
- Vascular pattern 8
- Vascular pattern 9
- Vascular pattern 10
- Vascular pattern 11

SUMMARY:
Retrospective analysis to the course and branching pattern as well as surgically relevant inner diameters and lengths of the superficial temporal artery (STA) by digital subtraction angiographies (DSA).

ELIGIBILITY:
Inclusion Criteria:

* good quality digital subtractions angiographies of the STA

Exclusion Criteria:

* bad quality digital subtractions angiographies of the STA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: clinic patients who underwent digital subtractions angiographie
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
vessel diameters | up to 36 month

SECONDARY OUTCOMES:
vessel length | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Hand, Plastic and Reconstructive Surgery with Burn Center BG Trauma Center, Tübingen, Germany

REFERENCES:
- [Background] Pinar YA, Govsa F. Anatomy of the superficial temporal artery and its branches: its importance for surgery. Surg Radiol Anat. 2006 Jun;28(3):248-53. doi: 10.1007/s00276-006-0094-z. Epub 2006 Mar 28. PMID 16568216